CLINICAL TRIAL: NCT00469079
Title: Comparing the Health Effects of Smokeless Tobacco, Cigarette Smoking, and New Tobacco Products Advertised as Safer Alternatives Part of Tobacco Exposure Reduction
Brief Title: Health Effects of SLT, Cigarette Smoking, and New Tobacco Products
Acronym: ANTS3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 010M79961; P50DA013333 (NIH)
Record Dates: First submitted 2007-05-03; First posted 2007-05-04 (Estimated); Results first posted 2014-04-14 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Nicotine Dependence
Keywords: Biomarkers; Smoking; Tobacco; Cessation
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Nicotine Chewing Gum; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Nicotine gum or nicotine lozenge; Dosage: 2 or 4 mg; Frequency: Daily; Duration: 5 weeks of use of which 1 week is tapering.
  Interventions: Drug: Nicotine gum and lozenge
- 2 (Experimental): Taboka - oral tobacco product Dosage: 0.84 to 1.26 mg free nicotine per g dry weight; Frequency: Daily; Duration: 5 weeks of use of which 1 week is tapering.
  Interventions: Other: Taboka
- 3 (Experimental): Camel Snus - oral tobacco product Dosage: 6.09 to 9.16 mg dry weight; Frequency: Daily; Duration: 5 weeks of use of which 1 week is tapering.
  Interventions: Other: Camel Snus

INTERVENTIONS:
Drug: Nicotine gum and lozenge — Nicotine replacement
  Other Names: Commit, Nicorette
  Arms: 1
Other: Taboka — smokeless tobacco product
  Arms: 2
Other: Camel Snus — smokeless tobacco product
  Arms: 3

SUMMARY:
The use of smokeless tobacco (ST) as a substitute for cigarette smoking has been suggested since it is considered by some to be a less harmful tobacco product (Russell, Jarvis and Feyerabend, 1980; Russell et al, 1981; Rodu, 1994). ST does not have the volatile constituents and carbon monoxide (CO) that are found in cigarette smoke. Since ST is not smoked there would be less risk of cardiovascular and lung disease. In addition the harm associated with second hand smoke would be eliminated. Although the health risks are reduced in ST users, they still exist due to the presence of nitrosamines found in ST. A better approach would be to use nicotine replacement that did not contain carcinogens, however the cost of such NRT could be prohibitive especially in third world countries where the rate of smoking is continuing to rise and the per capita income is much lower than in the United States.

Purpose: The goal of this study is to evaluate the health effects of Camel Snus, the new oral tobacco product produced by RJ Reynolds and Taboka, produced by Phillip Morris. These products are pasteurized rather than fermented and contain less moisture to eliminate spitting. They are marketed as an alternative to cigarette smoking.

DETAILED DESCRIPTION:
Cigarette smokers (n=125) will be recruited from the local metropolitan area using multiple media outlets. Subjects who are medically and psychologically healthy will be recruited for the study. Cigarette smokers will be informed of the study over the telephone and asked to answer a brief tobacco use history and medical screening questionnaire. If subjects pass the initial screening for the study, they will be asked to attend an orientation meeting at the Tobacco Use Research Center where the study will be explained in more detail, informed consent will be obtained and a full screening evaluation will occur. This evaluation includes the completion of several comprehensive tobacco use and social history forms and a complete physical and psychological screening.

Subjects will be required to attend the clinic once during Week 1 and once during Week 2 of the study in order to obtain baseline data. At the end of Week 2, cigarette smokers will be randomly assigned to either: 1) quit tobacco use and will be offered the choice of using nicotine gum or lozenge, depending on personal preference (n= 25) or they will be assigned to switch to: 2) Taboka (n=50) or 3) Camel Snus (n=50). Subjects sampled different flavors of the products for 1 week and then used the product for the next 4 weeks. During the four weeks, subjects will be asked to attend weekly clinic visits during which time study data will be collected. After the 4 weeks of study product use, subjects will be required to taper off of the tobacco or nicotine product over the next one week and then cease all tobacco use. Follow-up visits will be conducted 1 week and 11 weeks after completion of the study and outcome measures will be taken at that time. Blood and urine samples will be collected and analyzed for tobacco related toxicants during the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between 18-70 years of age
* Smoking at least 10 cigarettes/day for at least one year
* Good physical and mental health as evidenced by a medical history with no unstable medical conditions.

Exclusion Criteria:

* Uncontrolled chronic disease or condition that requires medical attention during the course of the study
* Contraindications for nicotine replacement products: active ulcers, recent heart attack, heart disease or irregular heart beat, uncontrolled high blood pressure, or medication use that might affect tobacco use
* Current unstable psychiatric diagnoses or persons who currently are adjusting medication dose. (within the last 3 months)
* Subjects with current or recent (within 6 months) alcohol or drug abuse problem
* Other regular tobacco use such as regular cigar or pipe smoking
* Currently using other nicotine replacement products
* Chronic use of any drug that could interact with the study drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2007-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, PHD, Principal Investigator — University of Minnesota
Locations (1):
- Tobacco Use Research Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Kotlyar M, Hertsgaard LA, Lindgren BR, Jensen JA, Carmella SG, Stepanov I, Murphy SE, Hecht SS, Hatsukami DK. Effect of oral snus and medicinal nicotine in smokers on toxicant exposure and withdrawal symptoms: a feasibility study. Cancer Epidemiol Biomarkers Prev. 2011 Jan;20(1):91-100. doi: 10.1158/1055-9965.EPI-10-0349. Epub 2010 Nov 10. PMID 21068204
- See also: Kotlyar M, Mendoza-Baumgart MI, Li ZZ, et al. Nicotine pharmacokinetics and subjective effects of three potential reduced exposure products, moist snuff and nicotine lozenge. Tob Control 2007;16:138-42. — http://www.ncbi.nlm.nih.gov/entrez/query.fcgi?cmd=Retrieve&db=PubMed&dopt=Citation&list_uids=17400953

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy smokers were recruited from the Twin Cities, MN metro area from November of 2006 through October of 2008.
Groups:
- Assigned to NRT: Nicotine gum or nicotine lozenge
- Assigned to Taboka: Taboka - oral tobacco product
- Assigned to Camel Snus: Camel Snus - oral tobacco product
Period: Overall Study
Arm/Group | Assigned to NRT | Assigned to Taboka | Assigned to Camel Snus
Started | 27 | 52 | 51
Completed | 18 | 30 | 32
Not Completed | 9 | 22 | 19
Not completed — Lack of Efficacy | 3 | 8 | 5
Not completed — Adverse Event | 1 | 3 | 2
Not completed — Lost to Follow-up | 4 | 8 | 10
Not completed — Withdrawal by Subject | 1 | 2 | 2
Not completed — Ineligible | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Assigned to NRT | Assigned to Taboka | Assigned to Camel Snus | Total
Number analyzed (Participants) | 27 | 52 | 51 | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 27 | 52 | 51 | 130
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (12.8) | 42.4 (11.2) | 43.6 (11.5) | 42.8 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 21 | 20 | 53
  Male | 15 | 31 | 31 | 77
Region of Enrollment [Number; unit: participants]
  United States | 27 | 52 | 51 | 130
Fagerstrom Test for Nicotine Dependence Score [Mean (Standard Deviation); unit: Scores on a scale] — Fagerstrom Test for Nicotine Dependence. Minimum value is 0 and maximum value is 10. Higher scores indicate greater dependence.
  Scores on a scale | 5.2 (1.2) | 3.8 (1.1) | 4.4 (1.6) | 4.5 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Toxicant Exposure by Products
Description: Levels of carcinogen biomarkers (NNAL) reported as difference between baseline and week 4 scores.
Time Frame: Baseline, 4 weeks
Population: All subjects who continued in the protocol were analyzed. Non-parametric Kruskal-Wallis method of analysis was used.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/ml
Groups:
- Medicinal Nicotine: 4 mg nicotine gum or nicotine lozenge
- Taboka: Taboka, a spitless oral tobacco product that has been discontinued. The product is pasteurized rather than fermented, leading to lower tobacco specific nitrosamine levels than conventional smokeless tobacco products.
- Snus: Camel Snus, a spitless oral tobacco product currently marketed as a substitute for cigarettes. The product is pasteurized rather than fermented, leading to lower tobacco specific nitrosamine levels than conventional smokeless tobacco products.
Arm/Group | Medicinal Nicotine | Taboka | Snus
Number analyzed (Participants) | 19 | 30 | 33
ng/ml
  Cotinine | 835.3 [351.5 to 1984.9] | 782.1 [414.5 to 1475.6] | 726.8 [333.7 to 1582.8]
  Total NNAL | 0.157 [0.096 to 0.255] | 0.281 [0.182 to 0.435] | 0.296 [0.191 to 0.458]
  Total NNN | 0.010 [0.003 to 0.034] | 0.011 [0.004 to 0.027] | 0.026 [0.012 to 0.057]
Statistical Analysis 1: Comparison: Medicinal Nicotine vs Taboka vs Snus; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis

2. Primary Outcome: Product Use at Week 4 of Intervention
Description: Self-reported daily use of the assigned study product. Range of scores is from 0 to about 20. Higher scores do not represent either a better or a worse outcome. Higher number of product used per day may indicate higher abuse liability of the product but may lead to a greater suppression in usual brand cigarette smoking. Lower number of product use per day may indicate lower abuse liability but may lead to lower suppression of usual brand smoking.
Time Frame: 4 weeks
Population: All subjects who completed intervention.
Measure: Least Squares Mean (Standard Error); unit: uses per day
Groups:
- Medicinal Nicotine: 4 mg nicotine gum or lozenge
- Taboka; Snus: A spitless, oral tobacco pouch.
Arm/Group | Medicinal Nicotine | Taboka | Snus
Number analyzed (Participants) | 18 | 30 | 32
uses per day | 7.27 (0.55) | 5.27 (0.42) | 6.76 (0.40)
Statistical Analysis 1: Comparison: Medicinal Nicotine vs Taboka vs Snus; Product use is by self-report and daily diaries; Test type: Superiority or Other; p = 0.05, Mixed Models Analysis

3. Primary Outcome: Abstinence From Tobacco at End of Treatment, 1 Week and 11 Weeks Post-intervention.
Description: This study was not powered to detect differences in smoking cessation rates between groups; however, smoking status was collected at each visit to obtain preliminary data. Point prevalence (no smoking during the previous 7 days) cigarette abstinence rates were calculated at the end of treatment and at each of the 2 follow-up visits (week 1 and 11 post-intervention). Continuous abstinence rates were calculated for the 4 week period between the week 1 and week 4 visits. Abstinence at all visits was assessed by self-report (i.e., no cigarettes smoked) and confirmed by an exhaled CO of less than 8 ppm. At the follow-up visits, abstinence was also confirmed by both exhaled CO concentrations and urinary cotinine concentration (<35 ng/mL).
Time Frame: 12 weeks
Population: Intent to treat model.
Measure: Number; unit: participants
Groups:
- Medicinal Nicotine: Nicotine gum or nicotine lozenge
- Taboka: Taboka - oral tobacco product
- Camel Snus: Camel Snus - oral tobacco product
Arm/Group | Medicinal Nicotine | Taboka | Camel Snus
Number analyzed (Participants) | 27 | 52 | 51
participants
  End of intervention continuous abstinence | 11 | 17 | 22
  1 week post-intervention point prevalence | 15 | 22 | 24
  11 weeks post intervention point prevalence | 9 | 12 | 16
Statistical Analysis 1: Comparison: Medicinal Nicotine vs Taboka vs Camel Snus; This study was not powered to detect differences in smoking cessation rates between groups; however, smoking status was collected to obtain preliminary data. Point prevalence (no smoking during the previous 7 days) cigarette abstinence rates were calculated at the week-4 visit and at each of the 2 follow-up visits. Continuous abstinence rates were calculated for the 4 week period between the week 1 and week 4 visits. Abstinence at all visits was assessed by self-report and confirmed by CO; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; A generalized linear mixed model was used for outcomes that had been repeatedly measured from baseline through the end of the treatment period; Other = 0

4. Secondary Outcome: Product Effect on Craving and Nicotine Withdrawal Symptoms at 1 Week.
Description: Changes in craving and withdrawal symptoms were assessed at the time of discontinuation of usual brand cigarettes (i.e., baseline compared to week 1). Assessments were made using the Minnesota Nicotine Withdrawal Scale, which measures abstinence effects from usual brand cigarettes. Total Score: Range of scores is from 0 to 28. All items with the exclusion of craving are summed. Craving Score: Range of score is from 0 to 4. A higher score would indicate more severe withdrawal.
Time Frame: Baseline and 1 week
Population: All subjects completing the intervention
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Medicinal Nicotine | Taboka | Snus
Number analyzed (Participants) | 18 | 30 | 32
units on a scale
  Craving Scores | 2.55 (0.18) | 2.76 (0.14) | 2.62 (0.13)
  Nicotine Withdrawal Scores | 8.15 (1.17) | 8.89 (0.86) | 8.61 (0.83)
Statistical Analysis 1: Comparison: Medicinal Nicotine vs Taboka vs Snus; A generalized linear mixed model was used for outcomes that had been repeatedly measured from baseline through the end of the treatment period. Each repeated-measures model included the treatment effect, a visit effect, the interaction between treatment and visit, the interaction between subject error and within-subject error terms; Test type: Superiority or Other; p > 0.10, Mixed Models Analysis; Mean difference between 3 groups = 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected during 4 weeks on study product.
Arm/Group | Assigned to NRT | Assigned to Taboka | Assigned to Camel Snus
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/52 | 0/51
Other Adverse Events (participants affected / at risk) | 18/27 | 28/52 | 39/51
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Assigned to NRT (N=27) | Assigned to Taboka (N=52) | Assigned to Camel Snus (N=51)
Dry Mouth (General disorders) | 4 (6) | 11 (16) | 13/27 (27)
Headaches (General disorders) | 6 (10) | 8 (8) | 7 (10)
Dizziness (Ear and labyrinth disorders) | 1 (1) | 6 (6) | 2 (2)
Lightheadedness (General disorders) | 2 (2) | 5 (5) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 10 (14) | 6 (11)
Stomach Aches (Gastrointestinal disorders) | 5 (6) | 5 (7) | 11 (14)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 5 (7)
Sore Jaw or Jaw Pain (General disorders) | 4 (7) | 1 (1) | 3 (4)
Shakiness (General disorders) | 1 (1) | 5 (6) | 1 (2)
Hiccups (General disorders) | 3 (7) | 3 (4) | 20 (35)
Sore Throat (General disorders) | 6 (8) | 3 (3) | 5 (10)
Mouth Sores (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (7) | 16 (27)
Sleep Disturbance (General disorders) | 8 (9) | 10 (12) | 11 (14)
Excessive Salivation (General disorders) | 4 (11) | 7 (9) | 15 (30)

LIMITATIONS AND CAVEATS:
Smokeless tobacco products commercially available have been introduced, withdrawn, or changed at a relatively rapid rate resulting in products that are no longer available and changes that occurred during the time period that the study occurred.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes